CLINICAL TRIAL: NCT05811260
Title: Effects of Myofascial Release Versus Post Facilitation Stretch Techniques on Pain,Range of Motion And Disability in Chronic Non Specific Low Back Pain.
Brief Title: MFR Versus PFS Techniques on Pain,Range of Motion And Disability in Chronic Non Specific Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0106
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Chronic Non Specific Low Back Pain
Keywords: Chronic pain,myofascial release technique, Postfacilitation stretch,Technique and low back pain.
MeSH Terms: conditions — Low Back Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Release (Active Comparator): Group A (Myofascial release technique) on low back 3 repetitions (30 second rest between reps), lasting for 30 s for each myofascial track for 1 set to targeted muscles (plantar fascia, gastrocnemius, hamstrings, and erector spinae). The position will be held for 10-15 seconds when a pain point is found lacrosse ball excellent for this type of massage because their surface area is much less than that of foam rollers.
  Interventions: Other: Myofascial Release technique
- Post facilitation stretch (Active Comparator): Group B (Post facilitation stretch) static stretching exercises for the low back (plantar fascia, gastrocnemius, hamstrings, and erector spinae). Static stretching involved 3 sets of 3 repetitions for each muscle with a 30-second hold and 30-second rest interval for each repetition.
  Interventions: Other: Post facilitation stretch .

INTERVENTIONS:
Other: Myofascial Release technique — on low back 3 repetitions (30 second rest between reps), lasting for 30 s for each myofascial track for 1 set to targeted muscles (plantar fascia, gastrocnemius, hamstrings, and erector spinae). The position will be held for 10-15 seconds when a pain point is found lacrosse ball excellent for this type of massage because their surface area is much less than that of foam rollers.
  Other Names: Myofascial Release technique for chronic non specific low back pain
  Arms: Myofascial Release
Other: Post facilitation stretch . — static stretching exercises for the low back (plantar fascia, gastrocnemius, hamstrings, and erector spinae). Static stretching involved 3 sets of 3 repetitions for each muscle with a 30-second hold and 30-second rest interval for each repetition.
  Other Names: Post facilitation stretch for chronic non specific low back pain.
  Arms: Post facilitation stretch

SUMMARY:
To compare effect of myofascial Release versus post facilitation stretch in term of pain ,range of motion and disability in chronic non specific low back pain in patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults already diagnosed with LBP
* Between ages group of 40-55 years.

Exclusion Criteria:

* Patients who had LBP originating from various pathologies, such as presence of
* cord compression,
* radiculopathy,
* osteoporosis,

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
. Numeric pain rating scale | 4 weeks
  NPRS is based on 11 points numerical rating scale for determining pain intensity, 0 ( no ;pain), 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Inclinometer | 4 weeks
  This instrument can measure Flexion, Extension, lateral flexion; a full range of tests ensures the best results. The Baseline Inclinometer is designed with your needs in mind; whether you need it for home or your professional clinic

OTHER OUTCOMES:
Modified Oswestry Disability index | 4 weeks
  Urdu version of Modified Oswestry Disability Index has become one of the principal condition specific outcome measures used in the management of spinal disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Study principal Investigator
Locations (1):
- DHQ, Layyah, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foster NE, Anema JR, Cherkin D, Chou R, Cohen SP, Gross DP, Ferreira PH, Fritz JM, Koes BW, Peul W, Turner JA, Maher CG; Lancet Low Back Pain Series Working Group. Prevention and treatment of low back pain: evidence, challenges, and promising directions. Lancet. 2018 Jun 9;391(10137):2368-2383. doi: 10.1016/S0140-6736(18)30489-6. Epub 2018 Mar 21. PMID 29573872
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870